CLINICAL TRIAL: NCT01119963
Title: 17-alpha-Hydroxyprogesterone Caproate (17P, Makena®) for Prolongation of Pregnancy in Women With Preterm Rupture of the Membranes (PROM), Double-blinded Randomized Clinical Trial
Brief Title: Progesterone (17P, Makena®) for Prolongation of Pregnancy in Women With Preterm Rupture of the Membranes (PROM)
Acronym: 17PinPROM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Organization: Pediatrix (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OBX0012
Record Dates: First submitted 2010-02-16; First posted 2010-05-10 (Estimated); Results first posted 2018-05-30 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Preterm Delivery
Keywords: Preterm delivery
MeSH Terms: conditions — Premature Birth | interventions — 17 alpha-Hydroxyprogesterone Caproate; Progesterone; Castor Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 17-alpha hydroxyprogesterone caproate, Makena® (Active Comparator): 250 mg of 17P, Makena® intramuscular (IM) weekly.
  Interventions: Drug: 17-alpha-hydroxy-progesterone caproate, Makena®
- Placebo (Placebo Comparator): Castor Oil (Placebo)intramuscular (IM) weekly
  Interventions: Drug: Castor Oil (Placebo)

INTERVENTIONS:
Drug: 17-alpha-hydroxy-progesterone caproate, Makena® — Intramuscular (IM) injection of 17P,Makena® (250mg) beginning as early as 23w0d administered weekly until 34w0d, documented fetal lung maturity at 32w0d - 33w6d, or delivery which ever comes first.
  Other Names: 17 alpha hydroxyprogesterone Caproate; 17P; 17Pc; 17HP; 170HP; 170HPC; Progesterone; Makena®
  Arms: 17-alpha hydroxyprogesterone caproate, Makena®
Drug: Castor Oil (Placebo) — IM injections of Placebo (castor oil) beginning as early as 23w0d administered weekly until 34w0d, documented fetal lung maturity at 32w0d - 33w6d, or delivery which ever comes first.
  Other Names: Placebo; Castor Oil
  Arms: Placebo

SUMMARY:
The objective of the study is to determine if a weekly dose of 17 hydroxyprogesterone caproate (17P, Makena®) given to women with preterm rupture of the membranes will:

1. increase the probability of continuing the pregnancy until a favorable gestational age.
2. increase the interval between randomization and delivery.
3. decrease neonatal morbidity.

DETAILED DESCRIPTION:
Preterm rupture of the membranes (PROM) is the leading identifiable cause of prematurity and accounts for about one-third of all preterm deliveries and 18-20% of perinatal deaths in the USA. When PROM occurs at very early gestational ages, the clinician must make a decision whether to attempt to prolong the pregnancy or whether to recommend prompt delivery. Both approaches carry substantial risk. The strategy of continuing the pregnancy is commonly called "expectant management." During expectant management, gestational age steadily increases, and the balance naturally shifts toward favoring delivery. Once the gestational age reaches 34 weeks, the risk of lethal or permanent sequelae of prematurity or minimal, so most clinicians agree that delivery is warranted. Despite an attempt at expectant management, the majority of patients with PROM will be delivered within the first week or so. Unfortunately, no intervention other than antibiotic prophylaxis or corticosteroids have been shown to prolong latency or reduce neonatal morbidity after PROM. Recent evidence suggests that prophylactic administration of progesterone medications may reduce the risk of preterm delivery in women with certain risk factors, notably those with a history of a prior preterm delivery and those with a shortened cervix discovered by ultrasound examination. Clearly, women with PROM are at very high risk of preterm delivery, so there is a pressing need to study whether 17 hydroxyprogesterone caproate (17P) is effective after PROM. Progesterone might be beneficial after PROM both because it tends to promote uterine quiescence by suppressing the formation of myometrial gap junctions and because it has anti-inflammatory properties, suppressing the production of inflammatory cytokines and thereby inhibiting cervical ripening. Inflammation is a major pathway leading to preterm labor, cervical dilation & preterm delivery. 17P would seem to be like an ideal candidate for prolongation of pregnancy after PROM.

This is a double-blinded, placebo-controlled, multicenter, randomized clinical trial of 17P versus placebo. The primary outcome measure will be the percentage of each group reaching either a gestational age of 34w0d or documentation of fetal lung maturity at 32w0d to 33w6d. Secondary outcomes will include the latency period for each group and the percentage of newborns in each group who have major neonatal morbidity or death.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 18 years old or older
2. Gestational Age (GA) 23w0d and 30w6d @ time of enrollment
3. Singleton pregnancy
4. PROM defined as either (a) or (b) or (c) below (a) Documentation of vaginal leakage of indigo carmine dye instilled via amniocentesis (b) Positive Amnisure® test (c) Two or more of (i) through (iv): i. Nitrazine test with pH of 7 or more ii. Positive fern test iii. Gross pooling of clear fluid iv. US exam showing oligohydramnios

Exclusion Criteria:

1. Any contraindication to expectant management
2. Any fetal condition likely to cause serious neonatal morbidity independent of gestational age
3. History of allergy to 17P
4. Any contraindications to 17P use (e.g. Thrombosis, Breast CA, abnormal vaginal bleeding unrelated to pregnancy, jaundice, liver disease, uncontrolled HTN)
5. Any medical condition currently treated with systemic steroid medications
6. Cervical cerclage present at the time of PROM
7. Informed consent not obtained.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Combs, MD, Principal Investigator — Obstetrix Medical Group
Locations (15):
- United States (15):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Desert Good Samaritan Hospital, Mesa, Arizona
  - Banner Good Samaritan Hospital, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Long Beach Memorial Medical Center, Long Beach, California
  - Good Samaritan Hospital, San Jose, California
  - OConnor Hospital, San Jose, California
  - Swedish Medical Center, Denver, Colorado
  - Presbyterian/St Luke's Hospital, Denver, Colorado
  - Norton Kosair Children's Hospital, Louisville, Kentucky
  - Spectrum Health Hospital, Grand Rapids, Michigan
  - Saint Luke's Hospital, Kansas City, Kansas City, Missouri
  - Sunrise Medical Center, Las Vegas, Nevada
  - University of Cincinnati, Cincinnati, Ohio
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Background] Amon E, Lewis SV, Sibai BM, Villar MA, Arheart KL. Ampicillin prophylaxis in preterm premature rupture of the membranes: a prospective randomized study. Am J Obstet Gynecol. 1988 Sep;159(3):539-43. doi: 10.1016/s0002-9378(88)80002-4. PMID 3421250
- [Background] Committee on Obstetric Practice.. ACOG committee opinion. Antenatal corticosteroid therapy for fetal maturation. American College of Obstetricians and Gynecologists. Int J Gynaecol Obstet. 2002 Jul;78(1):95-7. PMID 12197491
- [Background] ACOG Committee on Obstetric Practice. Use of progesterone to reduce preterm birth. ACOG Committee Opinion 291: 1-2, American College of Obstetricians and Gynecologists, 2003
- [Background] ACOG Committee on Practice Bulletins. Premature rupture of membranes. ACOG Practice Bulletin 80: 1-13, American College of Obstetricians and Gynecologists, 2007
- [Background] Ananth CV, Savitz DA, Williams MA. Placental abruption and its association with hypertension and prolonged rupture of membranes: a methodologic review and meta-analysis. Obstet Gynecol. 1996 Aug;88(2):309-18. doi: 10.1016/0029-7844(96)00088-9. PMID 8692522
- [Background] Armstrong J, Nageotte M for the Society for Maternal-Fetal Medicine. Can progesterone prevent preterm birth? Contemp Obstet Gynecol 2005 (Oct);30-43
- [Background] Bengtson JM, VanMarter LJ, Barss VA, Greene MF, Tuomala RE, Epstein MF. Pregnancy outcome after premature rupture of the membranes at or before 26 weeks' gestation. Obstet Gynecol. 1989 Jun;73(6):921-7. doi: 10.1097/00006250-198906000-00002. PMID 2726113
- [Background] Beydoun SN, Yasin SY. Premature rupture of the membranes before 28 weeks: conservative management. Am J Obstet Gynecol. 1986 Sep;155(3):471-9. doi: 10.1016/0002-9378(86)90257-7. PMID 3752169
- [Background] Caritis SN, Rouse DJ, Peaceman AM, Sciscione A, Momirova V, Spong CY, Iams JD, Wapner RJ, Varner M, Carpenter M, Lo J, Thorp J, Mercer BM, Sorokin Y, Harper M, Ramin S, Anderson G; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD), Maternal-Fetal Medicine Units Network (MFMU). Prevention of preterm birth in triplets using 17 alpha-hydroxyprogesterone caproate: a randomized controlled trial. Obstet Gynecol. 2009 Feb;113(2 Pt 1):285-92. doi: 10.1097/AOG.0b013e318193c677. PMID 19155896
- [Background] Caughey AB, Robinson JN, Norwitz ER. Contemporary diagnosis and management of preterm premature rupture of membranes. Rev Obstet Gynecol. 2008 Winter;1(1):11-22. PMID 18701929
- [Background] Combs CA, McCune M, Clark R, Fishman A. Aggressive tocolysis does not prolong pregnancy or reduce neonatal morbidity after preterm premature rupture of the membranes. Am J Obstet Gynecol. 2004 Jun;190(6):1723-8; discussion 1728-31. doi: 10.1016/j.ajog.2004.02.042. PMID 15284781
- [Derived] Combs CA, Garite TJ, Maurel K, Mallory K, Edwards RK, Lu G, Porreco R, Das A; Obstetrix Collaborative Research Network. 17-Hydroxyprogesterone caproate to prolong pregnancy after preterm rupture of the membranes: early termination of a double-blind, randomized clinical trial. BMC Res Notes. 2011 Dec 29;4:568. doi: 10.1186/1756-0500-4-568. PMID 22206581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants between the Gestational age of 23w0d-30w6d were approach in the hospital setting following confirmation of rupture of membranes.
Pre-assignment Details: We had two patient that consented to the study but were withdrawn prior to randomization because they began to go into labor
Period: Overall Study
Arm/Group | 17-alpha Hydroxyprogesterone Caproate, Makena® | Placebo
Started | 74 | 78
Completed | 73 | 77
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Age, Continuous
Groups:
- Total: Total of all reporting groups
Arm/Group | 17-alpha Hydroxyprogesterone Caproate, Makena® | Placebo | Total
Number analyzed (Participants) | 74 | 78 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (5.8) | 29.5 (5.7) | 29.7 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 78 | 152
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 16 | 37
  Not Hispanic or Latino | 53 | 61 | 114
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: this section does not include Hispanic or Latino so these numbers were removed from the total RACE section.
  Participants
    number analyzed (Participants) | 53 | 62 | 115
    American Indian or Alaska Native | 3 | 4 | 7
    Asian | 4 | 1 | 5
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 8 | 14 | 22
    White | 37 | 42 | 79
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 74 | 78 | 152
Marital Status [Count of Participants; unit: Participants]
  Married/Living with partner | 44 | 46 | 90
  Single/Widowed | 27 | 30 | 57
  Divorced/Separated | 3 | 0 | 3
  Other (Unknown) | 0 | 2 | 2
Education [Count of Participants; unit: Participants]
  < HS graduate | 6 | 10 | 16
  HS Graduate or equivalent | 11 | 18 | 29
  Some College | 22 | 15 | 37
  College Graduate | 17 | 15 | 32
  Not Reported | 18 | 20 | 38
Tobacco Use [Count of Participants; unit: Participants] | 4 | 5 | 9
Illicit Drug Use [Count of Participants; unit: Participants] | 7 | 14 | 21
Gestational Age at Membrane Rupture [Mean (Standard Deviation); unit: weeks] | 25.9 (3.0) | 26.6 (2.9) | 26.2 (3.0)
Gestational Age at time of randomization (wks) [Mean (Standard Deviation); unit: weeks] | 26.7 (2.5) | 27.1 (2.4) | 26.9 (2.5)
Gestational Age Stratum at randomization (wks) [Count of Participants; unit: Participants]
  23w0d-25w6d | 31 | 28 | 59
  26w0d - 28w6d | 24 | 27 | 51
  29w0d-30w6d | 19 | 23 | 42

OUTCOME MEASURES:

1. Primary Outcome: Gestational Age at Delivery
Description: Gestational age is measured in weeks, from the first day of the woman's last menstrual cycle to the date the baby was born.
Time Frame: Measured from day of last menstrual cycle to day of birth and measured in weeks.
Population: Intent to treat population (included all participants who were randomized, whether they received study medication or not).
Measure: Mean (Standard Deviation); unit: weeks.
Arm/Group | 17-alpha Hydroxyprogesterone Caproate, Makena® | Placebo
Number analyzed (Participants) | 73 | 77
weeks. | 29.2 (2.72) | 29.5 (2.74)

2. Secondary Outcome: Duration of Latency Period
Description: Secondary Outcomes:
  - Duration of latency period (time from randomization to birth)
Time Frame: average number of days measured from day of study entry until day of delivery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 17-alpha Hydroxyprogesterone Caproate, Makena® | Placebo
Number analyzed (Participants) | 73 | 77
days | 17.1 (16.08) | 17.0 (15.77)

ADVERSE EVENTS:
Time Frame: Up to 60 days post delivery or discharge which ever comes first
Groups:
- Neonate: 17-alpha Hydroxyprogesterone Caproate, Makena®: Neonate:
  250 mg of 17P, Makena® intramuscular (IM) weekly.
  17-alpha-hydroxy-progesterone caproate, Makena®: Intramuscular (IM) injection of 17P,Makena® (250mg) beginning as early as 23w0d administered weekly until 34w0d, documented fetal lung maturity at 32w0d - 33w6d, or delivery which ever comes first.
- Neonate: Placebo: Neonate:
  Castor Oil (Placebo)intramuscular (IM) weekly
  Castor Oil (Placebo): IM injections of Placebo (castor oil) beginning as early as 23w0d administered weekly until 34w0d, documented fetal lung maturity at 32w0d - 33w6d, or delivery which ever comes first.
Arm/Group | Neonate: 17-alpha Hydroxyprogesterone Caproate, Makena® | Neonate: Placebo | 17-alpha Hydroxyprogesterone Caproate, Makena® | Placebo
All-Cause Mortality (participants affected / at risk) | 3/73 | 2/77 | 0/73 | 0/77
Serious Adverse Events (participants affected / at risk) | 3/73 | 2/77 | 0/73 | 0/77
Other Adverse Events (participants affected / at risk) | 0/73 | 0/77 | 0/73 | 0/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neonate: 17-alpha Hydroxyprogesterone Caproate, Makena® (N=73) | Neonate: Placebo (N=77) | 17-alpha Hydroxyprogesterone Caproate, Makena® (N=73) | Placebo (N=77)
Congenital Diaphragmatic Hernia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — For all enrolled participants the number who had a newborn with a diagnosis of congenital diaphragmatic hernia noted at time of birth.
Respiratory Failure, Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — For all enrolled participants the number who had a newborn with a neonatal death in association with neonatal sepsis and respiratory failure events.
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — For all enrolled participants the number who had a newborn with a neonatal death following respiratory distress.
Atypical Pulmonary Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — For all enrolled participants the number who had a newborn with a neonatal deaths following a atypical pulmonary infection following birth
Suspected Pulmonary Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — For all enrolled participants the number who had a newborn death following suspected pulmonary hypertension.

LIMITATIONS AND CAVEATS:
One limitation is that we only studied one dose of 17OHPc (250mg) and only one frequency (once a week) however we did this to coincide with the study that showed benefits of 17OHPc in women with intact membranes with a history of preterm birth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No